CLINICAL TRIAL: NCT06000696
Title: Healthy At Home: Feasibility Trial of Home-Based Management of Patients with Chronic Obstructive Pulmonary Disease (COPD) Using Digital Technology
Brief Title: Healthy At Home Pilot
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: UMass Memorial Health (Other)
Responsible Party: Principal Investigator, Apurv Soni, Assistant Professor, University of Massachusetts, Worcester
Other Study IDs: 20224690
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: COPD; COPD Exacerbation; Emphysema or COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective is to conduct a pilot-feasibility trial of the "Healthy at Home" program, a multimodal intervention aimed at preventing acute care needs among COPD patients. The program will feature a digital platform and virtual pulmonary rehabilitation to facilitate complex care management of UMass Memorial Health Patients

DETAILED DESCRIPTION:
The Healthy at Home project is a pilot program aimed at improving care for patients who have COPD. This pilot aims to establish how self-management using a digital application, mobile health services, and support from a wellness coach can help achieve this goal. Participation in this study involves participants downloading a smartphone app, answering questionnaires, and wearing a Fitbit everyday, including during sleep throughout the 6-month study period. The investigators will ask that participants share their medical records and healthcare visit information through the secure study app, to help better understand how to treat patients with chronic health conditions. Participants will additionally have the option to enroll in Wellinks, a program that helps patients manage their breathing and COPD symptoms and provides patients with at-home medical equipment, one-on-one personalized virtual support from specially trained clinicians and coaches, and a separate easy-to-use app for tracking and communication.

ELIGIBILITY:
Inclusion Criteria:

* Receives healthcare through UMass Memorial Health
* Is at least 18 years old
* Has a self-reported or EMR observed diagnosis of COPD
* Has access to a smartphone (iPhone or Android) to download and use the study app(s)
* Lives within the geographic area served by the Mobile Integrated Health program

Exclusion Criteria:

* Lacks capacity to consent
* Does not understand English
* Does not have internet access on their smartphone at home
* Are currently enrolled in another investigational clinical trial
* Are or have previously been enrolled in any Wellinks program

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients of Umass Memorial Health system who have a diagnosis of COPD and live within the geographic area served by the Mobile Integrated Health program who are identified as potentially being a fit for the study program and are willing and able to download the study app and consent to the study via the app.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Enroll | 14 months
  Develop and use a smartphone app to enroll 100 UMass Memorial Health patients into the Healthy at Home program based on their short-term risk of requiring acute care needs.
Enhance | 18 months
  Enhance the existing Mobile Integrated Health (MIH) dashboard that currently only tracks care episodes by remotely collecting biometric data (oxygen saturation, respiratory rate, body temperature, heart rate) and participant reported data to allow the MIH paramedics to review longitudinal history of the patients prior to and after providing care.
Evaluate | 24 months
  Follow enrolled participants for six months to measure feasibility (adherence, usability) and clinical (patient-reported outcomes, healthcare utilization, total medical expenditure) outcomes at baseline, 3-months, and 6-months. Compare outcomes across full-intervention (Healthy at Home w/ virtual pulmonary therapy group), partial-intervention (Healthy at Home), and control (synthetic controls derived from EMR) after adjusting for baseline risk of acute-care needs.

CONTACTS AND LOCATIONS:
Overall Officials: Apurv Soni, MD, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connor L, Behar S, Tarrant S, Stamegna P, Pretz C, Wang B, Savage B, Scornavacca TT, Shirshac J, Wilkie T, Hyder M, Zai A, Toomey S, Mullen M, Fisher K, Tigas E, Wong S, McManus DD, Alper E, Lindenauer PK, Dickson E, Broach J, Kheterpal V, Soni A. Rationale and design of healthy at home for COPD: an integrated remote patient monitoring and virtual pulmonary rehabilitation pilot study. Pilot Feasibility Stud. 2024 Oct 28;10(1):131. doi: 10.1186/s40814-024-01560-x. PMID 39468649
- [Derived] O'Connor L, Behar S, Tarrant S, Stamegna P, Pretz C, Wang B, Savage B, Scornavacca T, Shirshac J, Wilkie T, Hyder M, Zai A, Toomey S, Mullen M, Fisher K, Tigas E, Wong S, McManus DD, Alper E, Lindenauer PK, Dickson E, Broach J, Kheterpal V, Soni A. Rationale and Design of Healthy at Home for COPD: an Integrated Remote Patient Monitoring and Virtual Pulmonary Rehabilitation Pilot Study. Res Sq [Preprint]. 2024 Apr 29:rs.3.rs-3901309. doi: 10.21203/rs.3.rs-3901309/v1. PMID 38746125